CLINICAL TRIAL: NCT04184518
Title: Phase II, Open-Label Study of Preliminary Efficacy of Durvalumab (MEDI4736) in Combination With Cediranib in Patients With Metastatic Uveal Melanoma
Brief Title: Durvalumab (MEDI4736) Plus Cediranib in Patients With Metastatic Uveal Melanoma
Acronym: CEDUVEAL-M
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The Cediranib producer laboratory decided to stop the development of this product.
Sponsor: Grupo Español Multidisciplinar de Melanoma (Other)
Collaborators: MFAR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM-1805; ESR-18-14002 (Other: AZ); 2019-001045-40 (EudraCT Number)
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Uveal Melanoma; Metastatic Cancer
Keywords: uveal melanoma; cediranib; durvalumab; liver metastasis
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis | interventions — cediranib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cediranib plus durvalumab (Experimental)
  Interventions: Drug: Cediranib Maleate; Drug: Durvalumab

INTERVENTIONS:
Drug: Cediranib Maleate — Cediranib 20mg, oral, 5 days on and 2 days off until disease progression
Drug: Durvalumab — Durvalumab 1500mg, intravenous, every 4 weeks until disease progression
  Other Names: MEDI4736

SUMMARY:
Phase II clinical trial aimed to evaluate the efficacy of the combination of cediranib and durvalumab in patients with metastatic uveal melanoma (mUM) with biopsiable disease at first line of after failure to first line systemic or liver directed therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed metastatic uveal melanoma with measurable disease not eligible for curative therapy.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. Patients must have at least 1 biopsiable liver metastasis.
* Patients can have received one prior therapy for metastatic disease, excepting for treatments listed in exclusion criteria.
* Patients must be 18 years of age or older at time of study entry.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
* Adequate normal organ and marrow function as defined below: Haemoglobin ≥9.0 g/dL, Absolute neutrophil count (ANC) > 1.5 x 109/L (> 1500 per mm3), Platelet count ≥ 100 x 109/L (>100,000 per mm3). Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with Coordinating Investigator. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) <2.5 x upper limit of normal (ULN) in the absence of liver metastases. If liver metastases are present, both AST and ALT must be no more than 5 x ULN. Creatinine clearance >30 ml/min calculated by Cockcroft-Gault or another validated method. Urine protein:creatinine ratio (UPC) ≤1 or ≤2+ proteinuria on 2 consecutive dipsticks taken no less than 1 week apart. Subjects with 2+ proteinuria on dipstick must also have UPC < 0.5 on 2 consecutive samples.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential as confirmed by a negative urine or serum pregnancy test within 7 days prior to inclusion. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply: Amenorrheic for ≥1 year in the absence of chemotherapy and/or hormonal treatments. Luteinizing hormone (LH) and/or follicle stimulating hormone and/or estradiol levels in the post-menopausal range. Radiation induced oophorectomy with last menses >1 year ago. Chemotherapy induced menopause with >1 year interval since last menses. Surgical sterilization (bilateral oophorectomy or hysterectomy) Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy). Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Must have a life expectancy of at least 12 weeks
* Subjects must be able to swallow and retain oral medications and be without clinically significant gastrointestinal illnesses that would preclude absorption of cediranib.
* Adequately controlled BP: Systolic BP ≤140 mmHg and diastolic BP ≤90 mmHg in the presence or absence of a stable regimen of antihypertensive therapy.

Exclusion Criteria:

* Patients with concomitant malignancy other than non-melanoma skin cancer, or superficial bladder cancer controlled with local treatment.
* Previous treatment with anti-angiogenic agents MEK, BRAF, ERK inhibitors.
* Previous treatment with anti-PD1/PDL1 (including durvalumab) treatments.
* Presence of brain or leptomeningeal involvement unless previously treated, off steroids at least 2 weeks, and considered stable. Patients with untreated central nervous system (CNS) metastases and/or carcinomatous meningitis identified either on the baseline brain imaging [RECIST]) obtained during the screening period or identified prior to signing the ICF. Patients whose brain metastases have been treated may participate provided they show radiographic stability (defined as 2 brain images, both of which are obtained after treatment to the brain metastases. These imaging scans should both be obtained at least four weeks apart and show no evidence of intracranial progression). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of ≤10mg/day of prednisone or its equivalent and anticonvulsants, for at least 14 days prior to the start of treatment. Brain metastases will not be recorded as RECIST Target Lesions at baseline.
* Patients weighing <30kg will be excluded from enrollment.
* Participation in another clinical study with an investigational product during the last 4 weeks.
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤28 days prior to the first dose of study drug If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by Sponsor designated Coordinating Investigator and Principal Investigator.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria: Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Coordinating Investigator. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Coordinating Investigator.
* Any concurrent chemotherapy, IMP, biologic, or hormonal therapy for cancer treatment different to cediranib and/or durvalumab. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
* Major surgery within a minimum of 2 weeks prior to inclusion; patients must have recovered from any effects of any major surgery prior to inclusion. Note: Local surgery of isolated lesions for palliative intent and minor surgeries performed to obtain biological material for the study (i.e. liver biopsy) are acceptable.
* History of allogeneic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion: Patients with vitiligo or alopecia. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement. Any chronic skin condition that does not require systemic therapy. Patients without active disease in the last 5 years may be included but only after consultation with the Coordinating Investigator. Patients with celiac disease controlled by diet alone.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, compromise cediranib absorption, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* History of another primary malignancy, except for: Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IMP and of low potential risk for recurrence. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease. Adequately treated carcinoma in situ without evidence of disease.
* History of active primary immunodeficiency.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion: Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection). Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IMP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IMP and up to 30 days after the last dose of IMP.
* Female patients who are pregnant (confirmed with positive pregnancy test) or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab and or cediranib therapy.
* History of severe allergic reaction attributed to cediranib or a similar VEGFR inhibitor or known hypersensitivity to any component of cediranib dose composition.
* Known allergy or hypersensitivity to durvalumab or any of the durvalumab excipients.
* History of gastrointestinal perforation. Subjects with a history of abdominal fistula will be eligible if: the fistula has been surgically repaired, there is no evidence of fistula for at least 6 months prior to inclusion, and the subject is deemed to be at low risk of recurrent fistula in the opinion of the Investigator.
* History of intra-abdominal abscess within 3 months prior to inclusion.
* Clinically significant signs and/or symptoms of bowel obstruction within 3 months prior to inclusion.
* Resting ECG with clinically significant abnormal findings. i.e. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).
* Subjects with any one or more of the following: History of myocardial infarction within 6 months prior to inclusion; patients with a history of myocardial infarction within 6 to 12 months prior to inclusion may be allowed following assessment. Unstable angina within 6 months prior to inclusion. Known significant cardiac disease (New York Heart Association [NYHA] classification of III or IV).
* Left ventricular ejection fraction < lower limit of normal (LLN) per institutional guidelines, or <55%, if threshold for normal is not otherwise specified by institutional guidelines, for patients with the following risk factors: Prior or planned treatment with anthracyclines (ie, PLD). Prior treatment with trastuzumab. Prior central thoracic radiation therapy (RT), including exposure of heart to therapeutic doses of ionizing RT. History of myocardial infarction within 6 to 12 months prior to inclusion. Prior history of other significant impaired cardiac function.
* History of stroke or transient ischemic attack within 6 months prior to inclusion.
* Evidence of any other disease, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that puts the subject at high risk for treatment-related complication.
* Prior enrollment or treatment in a previous durvalumab and/or cediranib clinical study regardless of treatment arm assignment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate by RECIST 1.1 | 24 months after start of treatment
  ORR calculated as the proportion of patient with a complete response (CR) or partial response (PR). The final statistical analysis of this endpoint is expected to be performed every 8 weeks since start of treatment.

SECONDARY OUTCOMES:
Median Progression-free survival (PFS) by RECIST 1.1 | 24 months after start of treatment
  Median time between start of treatment and date of progression of disease
Overall Survival Rate at 12 months | 12 months after start of treatment
  Proportion of patients alive 12 months since start of treatment
Overall Survival Rate at 24 months | 24 months after start of treatment
  Proportion of patients alive 24 months since start of treatment
Increase in effector CD8 T-cell response in the tumor induced by cediranib combined with durvalumab | 24 months after start of treatment
  Changes in the CD8 values from baseline
Number of participants with adverse events as assessed by CTCAE v5.0 | 24 months
Number of participants with serious adverse events as assessed by CTCAE v5.0 | 24 months
Number of participants with immune-related adverse events as assessed by CTCAE v5.0 | 24 months
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: José M. Piulats, Study Chair — Institut Català d'Oncología L'Hospitalet
Locations (5):
- Spain (5):
  - Instituto Catalá d'Oncología L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - H. U. Virgen de la Victoria, Málaga
  - Clínica Universidad de Navarra, Pamplona
  - H.U. Virgen Macarena, Seville
  - Hospital General Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided